CLINICAL TRIAL: NCT04836338
Title: Assessment of the GlideScope Spectrum Video Laryngoscope Blades and Stylet for Use in Neonate & Pre-Adolescent Populations: Pilot Manikin Study
Brief Title: GlideScope Spectrum Video Laryngoscope Blades and Stylet for Use in Neonate & Pre-Adolescent Populations
Status: Completed | Type: Observational
Sponsor: Verathon (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: GSX 1401
Record Dates: First submitted 2020-12-18; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Participants: Anesthesia and emergency medicine providers who perform pediatric orotracheal intubations
  Interventions: Device: orotracheal intubation

INTERVENTIONS:
Device: orotracheal intubation — orotracheal intubation

SUMMARY:
The overall purpose of this study is to assess the functionality & impact of the use of the newly designed GlideScope Spectrum pediatric video laryngoscope and stylet for the orotracheal intubation of neonates and pediatric patients, utilizing manikin models.

DETAILED DESCRIPTION:
The overall purpose of this study is to assess the functionality & impact of the use of the newly designed GlideScope Spectrum pediatric video laryngoscope blades and stylet for the orotracheal intubation of neonates and pediatric patients, utilizing manikin models. The hypothesis is that the Spectrum laryngoscope blades and stylet can improve the time and/or success of orotracheal intubation in a manikin.

Secondary aims of this study include assessing the impact of Spectrum pediatric video laryngoscope blades under simulated normal and difficult airway conditions on glottic view grade, mouth space, ease of blade insertion, ease of tracheal tube insertion, mechanisms of tracheal tube insertion impediment, and perceived overall clinical & functional usefulness in airways with predictors of difficult intubation.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia and emergency medicine providers who perform pediatric orotracheal intubations
* Able to give voluntary consent to participate in the study
* Are experienced with orotracheal intubation (> 50 times) using direct laryngoscopy or video laryngoscopy

Exclusion Criteria:

* Volunteers who are < 18 years of age
* Volunteers unable to read or understand English
* Unable to physically meet the demands of orotracheal intubation or those who have heart, wrist, or low back disease. Are not experienced with pediatric orotracheal intubations

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Clinicians, anesthesia, and emergency medicine providers who perform pediatric intubations. Participants will be recruited from Children's Medical Center, Dallas.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2016-02-09 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Time to intubate | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Time to intubate on each of 3 attempts per blade, on each manikin type.
First pass success rate | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  First pass success rate on each of 3 attempts per blade, on each manikin type. First pass success (FPS) is defined as the ability to place a tracheal tube below a patient's vocal cords on the first attempt without removing the video laryngoscope from the patient's mouth.
Overall performance and clinical utility using a 5-point Likert Scale | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Overall performance and clinical utility of single-use pediatric stylet; Using a 5-point LIKERT SCALE, participants will grade the following statements with regards to the use of the single-use pediatric stylet
  1. = strongly disagree
  2. = disagree
  3. = neutral
  4. = agree
  5. = strongly agree
     e.g. - Participants will assign a number to the following statements:
     * The pediatric style was easy to insert into the mouth of the when used with normal neonate manikin
     * The pediatric style was easy to insert into the mouth of the when used with the difficult neonate manikin
     * The pediatric style was easy to insert into the mouth of the when used with normal pediatric manikin

SECONDARY OUTCOMES:
Failed intubation attempt | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  The time taken for an intubation attempt that ultimately fails proper tube placement, or exceeds the allowed time for intubation under this protocol. Failed intubation attempt is defined as an attempt to intubate that does not result in tube placement, that is longer than 120 seconds, or results in a wrong placement of endotracheal tube (For example: Esophageal intubation, etc.).
Intubation success on first attempt | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Cumulative measure of intubation success on first attempt over 3 successive uses of the pediatric video laryngoscope, per blade, on each manikin type.

OTHER OUTCOMES:
Glottic view grade | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Glottic view grade on each of 3 attempts per blade, on each manikin type using the Cormack & Lehane grading scale:
  * Grade 1 = Full view of vocal cords
  * Grade 2a = Partial view of vocal cords
  * Grade 2b = Only arytenoids/posterior part of vocal cords
  * Grade 3 = Only epiglottis visible, no view of glottis or arytenoids
  * Grade 4 = Neither glottis nor epiglottis visible
Time to visualize glottis | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Time to visualize the glottis on each of 3 attempts per blade, on each manikin type.
Assessment of clinical utility and performance using a Lickert scale | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Assessment of the clinical utility and performance of the pediatric blades using a 5-point Lickert scale, where 1 = strongly disagree, 2 = disagree, 3= neutral, 4 = agree, 5 = strongly agree.
  * Ease of the pediatric video laryngoscope blade insertion when attempting to insert the pediatric video laryngoscope blade into manikin's mouth for each blade type and manikin type.
  * Ease of tracheal intubation when attempting to pass a tracheal tube below manikin's vocal cords using each of the pediatric video laryngoscope blades on each manikin type.
  * Assessment of the comfort of each blade handle during neonate/pediatric intubations.
  * Assessment of the blade and cable connection during neonate/pediatric intubation with each blade type.
  * Assessment of potential cable interference during neonate/pediatric intubation with each blade type.
Observational description of features causing impediments | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Participant self-reported observational description of potential features causing intubation impediments to tracheal tube insertion (e.g., tube hitting the epiglottis or tube hitting the arytenoid). Recorded by the study subject at the time of attempt at placing a tracheal tube below a patient's vocal cords using each of the pediatric video laryngoscope blades.
Overall clinical usefulness | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Recorded as excellent, good, fair, or inadequate by the study subject when using the pediatric video laryngoscope and stylet to place a tracheal tube below a patient's vocal cords.
Overall satisfaction of operator | 120 seconds - This is the maximum time allowed. After this time, it will be recorded as a failed attempt.
  Recorded as excellent, good, fair, or inadequate by the study subject when using each of the pediatric video laryngoscope blades and stylet to place a tracheal tube below manikin's vocal cords.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Olomu, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States